CLINICAL TRIAL: NCT05384340
Title: Nitrate-rich Beet Juice Intake and Aerobic Exercise on Cardiovascular Health of Postmenopausal Women With Arterial Hypertension
Brief Title: NO3-rich Beet Juice and Exercise on Postmenopausal Women Cardiovascular Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: BeetMPH5070
Record Dates: First submitted 2022-04-17; First posted 2022-05-20 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Arterial Hypertension; Postmenopausal; Menorrhagia; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Menorrhagia; Cardiovascular Diseases | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beet protocol (Experimental): Acute intervention: 1st day [140 ml - Beet It Juice, 800mg nitrate/day] Continued intervention: 2nd to 7th day [70 ml - Beet It Juice, 400mg nitrate/day] Exercise intervention [Treadmill - 40 minutes duration, 65% - 70% VO2 Peak]: Acute [Just on day] / Continued [First and latest day] Washout: 7 days
  Interventions: Dietary Supplement: Beetroot juice rich in nitrate
- Placebo protocol (Placebo Comparator): Acute intervention (1st day): [140 ml - Beet It Juice, 0mg nitrate/day] Continued intervention (2nd to 7th day): [70 ml - Beet It Juice, 0mg nitrate/day] Exercise intervention [Treadmill - 40 minutes duration, 65% - 70% VO2 Peak]: Acute [Just on day] / Continued [First and latest day] Washout: 7 days
  Interventions: Dietary Supplement: Beetroot juice rich in nitrate

INTERVENTIONS:
Dietary Supplement: Beetroot juice rich in nitrate — On the first day, an acute test will be carried out with beet juice rich in nitrate, in which two units of juice will be provided, totaling 140 ml (800 mg of nitrate) for each protocol. That is, each participant will receive 2 units of juice bottles. From the second to the seventh day, participants will receive 6 units of vials of the juice corresponding to the first intervention on the first visit to the laboratory and will drink one vial a day for a week. Of the 8 units (100%), six bottles (75%) will be provided for the participants to take home. On the seventh day of the intervention, the participants will return to the laboratory for the consumption of the seventh and last bottle of juice. Between one protocol and another, a 7-day washout interval will be given for the purification of the compounds provided by the protocols.

SUMMARY:
In the context of physical exercise, there is no evidence of the acute and continued use of beetroot juice with a previously recommended dose of nitrate (NO3) (>300mg) on the cardiovascular performance of hypertensive and postmenopausal women. We will investigate the effects of beetroot juice rich in NO3 acutely (first day: 140mL/800mg) and during a week with daily doses (second to the seventh day: 70mL/400mg) on blood pressure, heart rate (HR), cardiac autonomic control, EF, inflammatory, hormonal, and stress biomarkers oxidative stress and enzymes involved in nitric oxide synthesis and mitochondrial regulation, under resting conditions, as well as mediated by submaximal aerobic exercise sessions. Through a randomized, crossover, triple-blind, placebo-controlled clinical trial, 20 physically inactive hypertensive women will undergo an acute and 7-day trial, each with two intervention protocols: 1) placebo and 2) beetroot; in which will ingest beet juice with or without NO3 in its composition with a 7-day washout interval. On collection days, exercise will be performed on a treadmill for 40 minutes at a speed corresponding to 65-70% of VO2peak. The collection of variables (cardiovascular, autonomic, and blood samples for molecular analyses) of the study will take place at rest (120 minutes after ingestion of the intervention), during exercise (40 minutes), and in the effort recovery stage (during 65 minutes) based on previously validated protocols. The collections were arranged so that the measurement of one variable does not interfere with the other and that they have adequate intervals between them.

ELIGIBILITY:
Inclusion Criteria:

* Women with 50 to 65 old years;
* Physically inactive;
* Postmenopausal diagnosis (amenorrhea for 12 months or more);
* Arterial hypertension diagnosis (previously);
* Systolic blood pressure values >120mmHg up to 159mmHg and diastolic blood pressure values >80mmHg up to 99mmHg.

Exclusion Criteria:

* Previous history of acute myocardial infarction and/or stroke;
* Allergy or intolerance to nitrate, gluten, or milk;
* Medications (proton pump inhibitors, beta-blockers, calcium channels antagonists).

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Values of systolic and diastolic blood pressure (mmHg) | up to 2 years

SECONDARY OUTCOMES:
Values of heart rate variability (ms) | up to 2 years
Values of heart rate (beats per minute) | up to 2 years
Macrovascular function (Flow mediated dilatation%) | up to 2 years
Plasmatic concentrations of nitrate and nitrite (mmol/L) | up to 2 years
Blood concentration of Adiponectin (ug/mL) | up to 2 years
Blood concentration of Hormone-sensitive lipase (mmol/min per kg DM) | up to 2 years
Blood concentrations of C-reactive protein, Interleukin-6 and Interleukin-10 (ng/mL) | up to 2 years
Blood concentrations of Epinephrine and Norepinephrine (pg/mL) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bueno Júnior, PhD, Principal Investigator — EEFERP/USP
Locations (1):
- EEFERP - USP / Laboratório de Fisiologia do Exercício e Metabolismo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benjamim CJR, da Silva LSL, Sousa YBA, Rodrigues GDS, Pontes YMM, Rebelo MA, Goncalves LDS, Tavares SS, Guimaraes CS, da Silva Sobrinho AC, Tanus-Santos JE, Gualano B, Bueno Junior CR. Acute and short-term beetroot juice nitrate-rich ingestion enhances cardiovascular responses following aerobic exercise in postmenopausal women with arterial hypertension: A triple-blinded randomized controlled trial. Free Radic Biol Med. 2024 Feb 1;211:12-23. doi: 10.1016/j.freeradbiomed.2023.11.039. Epub 2023 Dec 11. PMID 38092272
- [Derived] Benjamim CJR, Sousa YBA, Porto AA, de Moraes Pontes YM, Tavares SS, da Silva Rodrigues G, da Silva LSL, da Silva Goncalves L, Guimaraes CS, Rebelo MA, da Silva Sobrinho AC, Tanus-Santos JE, Valenti VE, Gualano B, Bueno Junior CR. Nitrate-rich beet juice intake on cardiovascular performance in response to exercise in postmenopausal women with arterial hypertension: study protocol for a randomized controlled trial. Trials. 2023 Feb 7;24(1):94. doi: 10.1186/s13063-023-07117-2. PMID 36750904